CLINICAL TRIAL: NCT06712290
Title: Connective Tissue Matrix (CTM) Compared to Corticosteroid Injections: A Pilot Randomized Controlled Trial
Brief Title: Connective Tissue Matrix Compared to Steroid Injections for Rotator Cuff Tendinopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants met eligibility and the study was closed.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: CTM Biomedical (Industry)
Responsible Party: Principal Investigator, Sam Akhavan, MD, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-118
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Shoulder; Rotator cuff; Tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — Adrenal Cortex Hormones; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Corticosteroid (Placebo Comparator): Kenalog-40 is a long-acting corticosteroid injection for intramuscular (into the muscle) or intra-articular (into the joints) use. It may be used to treat many different types of inflammatory conditions.
  In this study, a 2.0cc dose injection of Kenalog-40 will be administered directly into the subacromial space using a 20G needle. 3mL of ropivacaine will be injected along with the steroid (as part of the same injection). Posttreatment pain control (hydrocodone/acetaminophen #20 5/500 mg) will be used.
  Interventions: Drug: Corticosteroid
- CTM Boost (Experimental): TM Boost (CTM Biomedical, Miami, FL) is a decellularized Human Cellular and Tissue Based Allograft (HCT/P) derived from placental connective tissue. It is marketed as an allograft for homologous use to supplement or replace damaged or inadequate connective tissue. It is regulated as a minimally-manipulated biologic by the FDA and is marketed as an allograft for homologous use to supplement or replace damaged or inadequate connective tissue. It is administered applied into the tissue via injection. Participant will undergo a single injection of 2.0cc of the injectable CTM allograft, administered using a 20G needle in the subacromial space. 3mL of ropivacaine will be mixed into the syringe prior to administration of the injection. Posttreatment pain control (hydrocodone/acetaminophen #20 5/500 mg) will be used.
  Interventions: Drug: celgene

INTERVENTIONS:
Drug: celgene — CTM Boost (CTM Biomedical, Miami, FL) is a decellularized Human Cellular and Tissue Based Allograft (HCT/P) derived from placental connective tissue. It is marketed as an allograft for homologous use to supplement or replace damaged or inadequate connective tissue. It is regulated as a minimally-manipulated biologic by the FDA and is marketed as an allograft for homologous use to supplement or replace damaged or inadequate connective tissue. It is administered applied into the tissue via injection.
  Participant will undergo a single injection of 2.0cc of the injectable CTM allograft, administered using a 20G needle in the subacromial space. 3mL of ropivacaine will be mixed into the syringe prior to administration of the injection. Posttreatment pain control (hydrocodone/acetaminophen #20 5/500 mg) will be used.
  Other Names: CTM boost
  Arms: CTM Boost
Drug: Corticosteroid — Kenalog-40 is a long-acting corticosteroid injection for intramuscular (into the muscle) or intra-articular (into the joints) use. It may be used to treat many different types of inflammatory conditions. In this study, a 2.0cc dose injection of Kenalog-40 will be administered directly into the subacromial space using a 20G needle. 3mL of ropivacaine will be injected along with the steroid (as part of the same injection). Posttreatment pain control (hydrocodone/acetaminophen #20 5/500 mg) will be used.
  Other Names: kenalog
  Arms: Corticosteroid

SUMMARY:
The goal of the study is to see which is better at treating patients which rotator cuff tendinopathy (RCT): a single injection of Connective Tissue Matrix boost (CTM) or a steroid shot.

Patients will be randomized (like flipping a coin) to the treatment. Patients and researchers will be blinded (not know) what group the patients are in.

Patients will come back to the study clinic at 6 weeks, 3 months and 6 months after the shot to answer questionnaires, have a physical exam, and complete physical function tests to check their shoulder.

DETAILED DESCRIPTION:
CTM vs. Steroid is a double-blind randomized controlled trial. Patients will be randomized to CTM Boost or Kenalog-40 (corticosteroid). Patients will be followed for six months and have three follow-up visits where they will have a physical exam, complete questionnaires, have a physical exam, including physical functional assessments, be screened for adverse events. Data will be collected from their medical chart after each visit.

CTM Boost (CTM Biomedical, Miami, FL) is a tissue allograft derived from decellularized, particulate human placental connective tissue. It is regulated as a minimally-manipulated human cell, tissue, and cellular and tissue-based product (HCT/P) biologic by the FDA and is marketed for homologous use to supplement or replace damaged or inadequate connective tissue. It is implanted via injection into the tissue. CTM Boost is available in a range of volumes. In this study, the 2.0cc volume of CTM Boost will be administered by injection directly into the subacromial space using a 20G needle.

Kenalog-40 is a long-acting corticosteroid injection for intramuscular (into the muscle) or intra-articular (into the joints) use. It may be used to treat many different types of inflammatory conditions. In this study, a 2.0cc dose injection of kenalog-40 will be administered directly into the subacromial space using a 20G needle (for patients randomized to this control arm).

Study Questionnaires are as follows:

* WORC: The WORC has 21 items in four domains, including physical symptoms (10 questions), sports/recreation/work (4 questions), lifestyle (4 questions) and emotions (3 questions). Raw scores range from 0 to 2100, with a higher score indicating decreased quality of life because of pathological condition of the rotator cuff.
* SANE: The Single Assessment Numeric Evaluation (SANE) is a patient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline. SANE scores are most commonly used by orthopedic sports specialist surgeons, and usually for the shoulder and the knee.
* VAS: The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 (no pain) and 10 (pain as bad as it could possibly be).
* ASES: The ASES score is a 10-item measure of shoulder pain and function. Pain is assessed on a 10-cm visual analog scale (VAS) and accounts for 50% of the total score. The remaining 50% of the score is determined by the responses to 10 4-point Likert-scale questions related to physical function
* Functional Assessments: various arm/shoulder exercises with dumbbells, weights or resistance. Time until patient is fatigued and/or number of repetitions will be measured.

  * These tests will include the following:

    * Empty can exercise with dumbbell resistance: Arm held in a position with weighted resistance, while measuring number of seconds to fatigue (or unable to maintain arm at 90 degrees).
    * Side-lying external rotation with dumbbell resistance: Lie on side (opposite shoulder) with weight held in hand, elbow flexed to 90 degrees while rotate through a full range of motion at the shoulder. The number of repetitions during a 30-second period are recorded.

Full can exercise with dumbbell resistance: Stand parallel to wall with the handheld in a fist and shoulder forward flexed parallel to the floor. A measuring stick will be used to measure how far forward on the yardstick patient can reach. The number of repetitions during a 60-second period are recorded.

External rotation of shoulder at 0 and 90 degrees with Thera-Band resistance. Patient will be instructed to perform rapid swinging motions in a 30-degree arc until fatigued.

Safety Evaluation:

* Infection
* Tear of the tendon
* Shoulder stiffness
* Admission to the hospital for a shoulder-related issue
* Surgical rotator cuff repair or subacromial decompression.

Data collected from a medical record review:

MRN Age Gender Weight Height Comorbidities Duration of symptoms Smoking status Diabetes Shoulder imaging reports from pre-enrollment MRI/xray Progress/Office notes Concomitant Medication

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old with rotator cuff tendinopathy
* A corticosteroid or CTM-type injection was determined by the clinician to be the proper medical treatment course and patient is willing to undergo the injection

Exclusion Criteria:

* Patients with adhesive capsulitis
* Patients with acromio-clavicular joint impingement, retracted tears, significant labral lesions or significant glenohumeral arthrosis
* Patients with joint instability
* History of shoulder surgery or corticosteroid injection in the past 3 months
* Patients with a history of chronic steroid treatment for any medical reason
* Patients with medical conditions that may affect healing, such as

  * End-stage renal disease
  * Uncontrolled diabetes
  * Peripheral vascular disease
  * Severe and/or systemic immunocompromising conditions such as Lupus or HIV infection
* Patients who are pregnant or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Raw WORC Score at 3 Month Visit | 3 Month Visit
  The primary outcome will be raw WORC score at the Month 3 visit. WORC is a patient-reported quality of life outcome measure for patients with rotator cuff disorders. The raw score obtained from scoring a completed questionnaire ranges from 0 to 2100, where higher scores indicate poorer quality of life.

SECONDARY OUTCOMES:
WORC Score | Baseline, Week 6, Month 3, Month 6 Visits
  WORC: The WORC has 21 items in four domains, including physical symptoms (10 questions), sports/recreation/work (4 questions), lifestyle (4 questions) and emotions (3 questions). Raw scores range from 0 to 2100, with a higher score indicating decreased quality of life because of pathological condition of the rotator cuff.
VAS: The Visual Analogue Scale | Baseline, Week 6, Month 3, Month 6 Visits
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
SANE: The Single Assessment Numeric Evaluation | Baseline, Week 6, Month 3, Month 6 Visits
  The SANEpatient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline. SANE scores are most commonly used by orthopedic sports specialist surgeons, and usually for the shoulder and the knee.
ASES | Baseline, Week 6, Month 3, Month 6 Visits
  The ASES score is a 10-item measure of shoulder pain and function. Pain is assessed on a 10-cm visual analog scale (VAS) and accounts for 50% of the total score. The remaining 50% of the score is determined by the responses to 10 4-point Likert-scale questions related to physical function
Functional Assessments: Empty can exercise | Baseline, Week 6, Month 3, Month 6 Visits
  Empty can exercise with dumbbell resistance: Arm held in a position with weighted resistance, while measuring number of seconds to fatigue (or unable to maintain arm at 90 degrees). Time until patient is fatigued
Functional Assessments: External Rotation with Dumbell | Baseline, Week 6, Month 3, Month 6 Visits
  Side-lying external rotation with dumbbell resistance: Lie on side (opposite shoulder) with weight held in hand, elbow flexed to 90 degrees while rotate through a full range of motion at the shoulder. The number of repetitions during a 30-second period are recorded.
Functional Assessments: Full can exercise with dumbbell resistance | Baseline, Week 6, Month 3, Month 6 Visits
  Stand parallel to wall with the handheld in a fist and shoulder forward flexed parallel to the floor. A measuring stick will be used to measure how far forward on the yardstick patient can reach. The number of repetitions during a 60-second period are recorded.
Functional Assessments: External rotation of shoulder at 0 and 90 degrees with Thera-Band resistance | Baseline, Week 6, Month 3, Month 6 Visits
  Patient will be instructed to perform rapid swinging motions in a 30-degree arc until fatigued.
Safety Evaluations; Adverse Events; Serious Adverse Events | Week 6, Month 3, Month 6 Visits
  * Infection
  * Tear of the tendon
  * Shoulder stiffness
  * Admission to the hospital for a shoulder-related issue
  * Surgical rotator cuff repair or subacromial decompression.

CONTACTS AND LOCATIONS:
Locations (1):
- Allegheny Health Network Federal North Medical Office Building, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Braun C, Handoll HH. Estimating the Minimal Important Difference for the Western Ontario Rotator Cuff Index (WORC) in adults with shoulder pain associated with partial-thickness rotator cuff tears. Musculoskelet Sci Pract. 2018 Jun;35:30-33. doi: 10.1016/j.msksp.2018.02.003. Epub 2018 Feb 12. PMID 29471221
- [Result] Chen J, Svensson J, Sundberg CJ, Ahmed AS, Ackermann PW. FGF gene expression in injured tendons as a prognostic biomarker of 1-year patient outcome after Achilles tendon repair. J Exp Orthop. 2021 Mar 11;8(1):20. doi: 10.1186/s40634-021-00335-0. PMID 33694106
- [Result] Dean BJ, Snelling SJ, Dakin SG, Murphy RJ, Javaid MK, Carr AJ. Differences in glutamate receptors and inflammatory cell numbers are associated with the resolution of pain in human rotator cuff tendinopathy. Arthritis Res Ther. 2015 Jul 10;17(1):176. doi: 10.1186/s13075-015-0691-5. PMID 26160609
- [Result] Giovannetti de Sanctis E, Franceschetti E, De Dona F, Palumbo A, Paciotti M, Franceschi F. The Efficacy of Injections for Partial Rotator Cuff Tears: A Systematic Review. J Clin Med. 2020 Dec 25;10(1):51. doi: 10.3390/jcm10010051. PMID 33375716